CLINICAL TRIAL: NCT05148052
Title: Effect of Upper Extremity Rehabilitation Using Fully-immersive Virtual Reality for Motor Recovery in Chronic Stroke Patients: A Prospective, Multicenter, Single-blind, Explorative, Randomized Crossover Trial
Brief Title: Effect of Upper Extremity Rehabilitation Using Immersive Virtual Reality in Chronic Stroke Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); National Traffic Injury Rehabilitation Hospital (Unknown); Korea Workers' Compensation and Welfare Service Incheon Hospital (Unknown)
Responsible Party: Principal Investigator, Han Gil Seo, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Stroke-VR-U/Ex
Record Dates: First submitted 2021-11-12; First posted 2021-12-08 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke; Virtual reality; Upper Extremity Paresis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional therapy first (Experimental): Group receiving conventional occupational therapy first and then virtual reality exergames.
  Interventions: Device: Virtual reality exergames; Behavioral: Conventional occupational therapy
- Virtual reality first (Experimental): Group receiving virtual reality exergames with virtual reality first and then conventional occupational therapy.
  Interventions: Device: Virtual reality exergames; Behavioral: Conventional occupational therapy

INTERVENTIONS:
Device: Virtual reality exergames — Twelve sessions of virtual reality exergames involving upper extremities will be conducted. Each session is 30 minutes and will be held 3 times a week. The washout period between the two types of interventions is 2 weeks.
Behavioral: Conventional occupational therapy — Conventional occupational therapy involving upper extremities will be conducted. Each session is 30 minutes and will be held 3 times a week. The washout period between the two types of interventions is 2 weeks.

SUMMARY:
The study aimed to investigate the effect of exergames using virtual reality with head mounted device on motor recovery of upper extremities in chronic stroke patients.

DETAILED DESCRIPTION:
This is a crossover study for comparing conventional occupational therapy and exercise with game format using virtual reality (virtual reality exergame). The virtual reality exergame is designed to maximize the movement of upper extremities, primary to the shoulder and elbow. Fifteen chronic stroke patient will receive conventional occupational treatment and virtual reality exergame in random order with a two-week-washout period. Outcome measures will be evaluated within two days before and after each treatment, conventional treatment and virtual reality exergame.

*Due to recruitment challenges, the anticipated enrollment has been revised from 36 to 15.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients who have passed 6 months or more without additional stroke after the first stroke
* Patients with upper extremity dysfunction due to stroke (ischemic, hemorrhagic)
* Patients who can move the upper extremity against gravity with a manual muscle test of grade 3 or higher in the affected shoulder and elbow, respectively
* Patients who can stably maintain a sitting position
* Patients who voluntarily agreed to participate in the study

Exclusion Criteria:

* Patients with moderate or severe cognitive impairment with a score of 18 or less on the Mini-Mental Status Examination (K-MMSE)
* Patients with other causes of upper extremity dysfunction, such as peripheral nerve damage, joint disease, etc.
* Patients with a history of severe vertigo or epilepsy
* Patients with medical reasons such as medical conditions that make it difficult to participate in research
* Patients who may be pregnant or who are pregnant or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test | Within 2 days after the end of each intervention
  As an upper extremity function evaluation tool, it tests grasp, grip, pinch, and gross arm movement function as sub-tests.

SECONDARY OUTCOMES:
Box and Block test | Within 2 days after the end of each intervention
  an upper extremity function evaluation tool
Fugl-Meyer (FM) Assessment | Within 2 days after the end of each intervention
  an upper extremity function evaluation tool
Modified Barthel Index | Within 2 days after the end of each intervention
  an evaluation tool for assessing activities of daily living
Grip strength | Within 2 days after the end of each intervention
  Strength of hand grip, palmar pinch and lateral pinch power measured by grip force meter
Beck Depression Inventory (BDI) | Within 2 days after the end of each intervention
  an evaluation tool for severity of depression in normal and psychiatric populations
Simulator Sickness Questionnaire | Day 1 and Day 12 of virtual reality exergames intervention
  an evaluation tool for assessing the subjective severity of simulator sickness symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Han Gil Seo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - National Traffic Injury Rehabilitation Hospital, Yangp'yŏng, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul